CLINICAL TRIAL: NCT07072403
Title: Safety and Efficacy of Trametinib for Complicated Vascular Anomalies: A Multicenter Prospective Study
Brief Title: Trametinib Treatment for Complicated Vascular Anomalies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCT20250701
Record Dates: First submitted 2025-07-07; First posted 2025-07-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Vascular Anomalies
Keywords: complicated vascular anomalies
MeSH Terms: conditions — Vascular Malformations | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Trametinib (Experimental): Patients will receive oral trametinib once daily
  Interventions: Drug: Trametinib tablet

INTERVENTIONS:
Drug: Trametinib tablet — Drug is supplied in 0.5 mg and 2 mg tablets

SUMMARY:
Complicated vascular anomalies have diverse etiologies and variable clinical manifestations, and no standardized treatment protocol has been established. Since most patients present with diffuse lesions that are difficult to resect surgically, identifying effective therapeutic strategies is of critical importance. This study aims to evaluate the safety and efficacy of systemic trametinib therapy in patients with complicated vascular anomalies.

DETAILED DESCRIPTION:
In recent years, with the widespread application of molecular diagnostic technologies and the growing awareness of complicated vascular anomalies among clinicians, an increasing number of molecular alterations have been identified in these disorders. This progress has brought new hope for patients who previously lacked standardized treatment options. Multiple somatic point mutations have been discovered in complicated vascular anomalies, and case reports have demonstrated significant therapeutic benefits from mutation-based targeted therapies-particularly in patients with NRAS mutations treated with MEK inhibitors. However, to date, there have been no prospective studies evaluating the safety and efficacy of trametinib in pediatric patients with complicated vascular anomalies. Such research is urgently needed to provide robust clinical evidence to guide treatment decisions for this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

* -Presenting a complicated vascular anomalies vascular anomalies with the following characteristics:

  1. Male and female;
  2. Between 1 and 18 years of age;
  3. Complicated vascular anomalies vascular anomalies diagnosis was confirmed by local investigators and by consensus of our multidisciplinary vascular anomaly group at the West China Hospital of Sichuan University based on:

Biopsy; Compatible MRI findings; History and clinical features.

Exclusion Criteria:

1. Patients have allergy or contraindication to MEK inhibitor
2. Exposure to chemotherapy, embolization, corticosteroids, propranolol, sclerotherapy or any other investigational agents within 1 weeks before enrolment on study;
3. Patients had a history of a major surgery within 2 weeks before enrollment;
4. Any known evidence of significant local or systemic uncontrolled infection, defined as receiving intravenous antibiotics at the time of enrollment;
5. Impairment of gastrointestinal function or chronic gastrointestinal disease that may significantly alter the absorption of trametinib.
6. Concurrent severe and/or uncontrolled medical diseases that could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
7. Patients with inadequate liver function:

   Total bilirubin higher than or equal to 1.5 × the upper limit of the normal (ULN) for age and alanine aminotransferase and aspartate aminotransferase higher than or equal to 2.5 × the ULN for age.
8. Patients with inadequate renal function:

   0-5 years of age maximum serum creatinine (mg/dL) of 0.8; 6-10 years of age maximum serum creatinine (mg/dL) of 1.0; 11-14 years of age maximum serum creatinine (mg/dL) of 1.2;
9. Adequate bone marrow function:

   Absolute neutrophil count lower than 1 × 109/L;
10. History of a malignancy within 5 years;
11. HIV infection or known immunodeficiency;
12. Patients with an inability to participate in or follow-up during the study treatment and assessment plan;
13. Inability to give informed consent.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving an objective response at month 12 | 12 months
  Objective response was defined as ≥20% reduction in lesion volume compared to that at baseline.

SECONDARY OUTCOMES:
The proportion of patients achieving an objective response at month 6 | 6 months
  Objective response was defined as ≥20% reduction in lesion volume compared to that at baseline.
lesion responses | 6 and 12 months
  The primary endpoint was classified as follow: -Complete involution: 100% resolution of the measured lesion volume; -Nearly complete involution was defined as decrease of ≥75% and <100%; -Partial involution was defined as decrease of ≥20% and <75%; -No change was defined as <20% increase and <20% decrease in the volumes of LM lesions; -Further growth was defined as ≥20% increase in the volume of index compared with the baseline volume measured. Lesion responses were overall lesion response rate and good lesion response rate. Overall lesion response comprised complete, nearly complete and partial involutions. Good lesion response comprised complete and nearly complete involutions.
Quality of life (QOL) in patients | 12 months
  Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Infant Scales (<2 years) or Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Scales (2-18 years) were used.
Disease sequelae | 12 months
  Disease sequelae were assessed by site investigators at month 12. The site investigators assessed patients' extremity swelling (if any), general physical activity and exercise levels.
Frequency of adverse events | 12 months
  Frequency of adverse events (e.g. gastrointestinal disorders, blood and lymphatic system disorders, metabolic disorders or other abnormal laboratory results, skin disorders and general disorders, etc.) collected by investigator and reported by parents. All adverse events were collected and graded according to Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0). The causality of the adverse event was determined by the multidisciplinary staff and was classified as definitively not related, probably not related, possibly related, probably related, or definitively related. Any dose reductions, interruptions, or cessations enacted at the discretion of the investigators were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Croteau SE, Kozakewich HP, Perez-Atayde AR, Fishman SJ, Alomari AI, Chaudry G, Mulliken JB, Trenor CC 3rd. Kaposiform lymphangiomatosis: a distinct aggressive lymphatic anomaly. J Pediatr. 2014 Feb;164(2):383-8. doi: 10.1016/j.jpeds.2013.10.013. Epub 2013 Nov 16. PMID 24252784
- [Background] Zhou Z, Qiu T, Zhou J, Zhang Z, Gong X, Zhang X, Lan Y, Yang C, Zhang Y, Xiang S, Ji Y. Clinical features and current management experience in Gorham-Stout disease: a systematic review. Orphanet J Rare Dis. 2025 Mar 19;20(1):134. doi: 10.1186/s13023-025-03649-9. PMID 40102890
- [Background] Foster JB, Li D, March ME, Sheppard SE, Adams DM, Hakonarson H, Dori Y. Kaposiform lymphangiomatosis effectively treated with MEK inhibition. EMBO Mol Med. 2020 Oct 7;12(10):e12324. doi: 10.15252/emmm.202012324. Epub 2020 Sep 7. PMID 32894644
- [Background] Li D, Sheppard SE, March ME, Battig MR, Surrey LF, Srinivasan AS, Matsuoka LS, Tian L, Wang F, Seiler C, Dayneka J, Borst AJ, Matos MC, Paulissen SM, Krishnamurthy G, Nriagu B, Sikder T, Casey M, Williams L, Rangu S, O'Connor N, Thomas A, Pinto E, Hou C, Nguyen K, Pellegrino da Silva R, Chehimi SN, Kao C, Biroc L, Britt AD, Queenan M, Reid JR, Napoli JA, Low DM, Vatsky S, Treat J, Smith CL, Cahill AM, Snyder KM, Adams DM, Dori Y, Hakonarson H. Genomic profiling informs diagnoses and treatment in vascular anomalies. Nat Med. 2023 Jun;29(6):1530-1539. doi: 10.1038/s41591-023-02364-x. Epub 2023 Jun 1. PMID 37264205
- [Background] Barclay SF, Inman KW, Luks VL, McIntyre JB, Al-Ibraheemi A, Church AJ, Perez-Atayde AR, Mangray S, Jeng M, Kreimer SR, Walker L, Fishman SJ, Alomari AI, Chaudry G, Trenor Iii CC, Adams D, Kozakewich HPW, Kurek KC. A somatic activating NRAS variant associated with kaposiform lymphangiomatosis. Genet Med. 2019 Jul;21(7):1517-1524. doi: 10.1038/s41436-018-0390-0. Epub 2018 Dec 13. PMID 30542204